CLINICAL TRIAL: NCT00623597
Title: A Phase I/II Study of Invirase® Boosted With Ritonavir in HIV Infected Infants and Children 4 Months to Less Than 6 Years Old
Brief Title: A Study of Invirase (Saquinavir)/Ritonavir in HIV-Infected Infants and Children.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV20911; 2007-004617-34
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ritonavir; Drug: saquinavir [Invirase]

INTERVENTIONS:
Drug: ritonavir — 2.5-3.0mg/kg po bid (starting dose) for 48 weeks
Drug: saquinavir [Invirase] — 50mg/kg po bid (starting dose) for 48 weeks

SUMMARY:
This single arm study will assess the pharmacokinetics, safety and activity of saquinavir (Invirase hard gel capsules, film coated tablets or opened capsules) boosted by combination with ritonavir, in HIV-1 infected infants and children between the ages of 4 months and 6 years. Patients will commence treatment with saquinavir 50mg/kg bid plus ritonavir 2.5mg/kg or 3.0mg/kg (dependent on body weight), and a background antiretroviral regimen. If drug exposures are found to be dissimilar to those previously seen in older children and adults, or are associated with toxicities, subsequent dose adjustments will be made. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* infants and children, 4 months to <6 years;
* confirmed HIV-1 infection;
* patients for whom saquinavir/ritonavir together with >=2 background ARVs is considered appropriate.

Exclusion Criteria:

* body weight >4kg/8.8 pounds;
* use of any concomitant medications that may interfere with the pharmacokinetics of saquinavir or ritonavir;
* malabsorption, severe chronic diarrhea or vomiting within 28 days of the study.

Ages: 4 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Argentina (2):
  - Buenos Aires
  - Santa Fe
- Spain (2):
  - Madrid, Madrid
  - Valencia, Valencia
- Thailand (4):
  - Bangkok
  - Khon Kaen
  - Pathumwan
  - Payathai

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 18 participants were recruited from 8 centers in Argentina (3 centers), Spain (1 center) and Thailand (4 centers). This study was conducted between May 20, 2008 and March 11, 2010.
Pre-assignment Details: Participants were human immunodeficiency virus (HIV) infected infants and young children who met the eligibility criteria were stratified into 2 groups - low age (>= 4 months to <2 years) and high age group (>= 2 years to <6 years). Participants commenced treatment with saquinavir and ritonavir along with background antiretroviral (ARV) regimen.
Groups:
- Group A: Participants (infants >= 4 months to <2 years old) received saquinavir at a dose of 50 milligram per kilogram (mg/Kg) twice a day (BID) and ritonavir at a dose of 3 mg/kg BID for body weight from 5 to < 15 kg, 2.5 mg/kg BID for body weight from 15 to 40 kg and 100 mg BID for body weight > 40 kg plus >= 2 background ARVs. After 14 days of treatment (or Day 28 for participants switching from an NNRTI containing regimen), saquinavir and ritonavir dose adjustments were made within the age group or for individual participants as deemed appropriate. The highest dose for saquinavir/ritonavir that was to be administered was not to exceed 1000 mg/100 mg BID. Participants received treatment for 48 weeks.
- Group B: Participants (children >= 2 years to <6 years old) received saquinavir at a dose of 50 mg/Kg BID and ritonavir at a dose of 3 mg/kg BID for body weight from 5 to < 15 kg, 2.5 mg/kg BID for body weight from 15 to 40 kg and 100 mg BID for body weight > 40 kg plus >= 2 background ARVs. After 14 days of treatment (or Day 28 for participants switching from an NNRTI containing regimen), saquinavir and ritonavir dose adjustments were made within the age group or for individual participants as deemed appropriate. The highest dose for saquinavir/ritonavir that was to be administered was not to exceed 1000 mg/100 mg BID. Participants received treatment for 48 weeks.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 5 | 13
Completed | 4 | 13
Not Completed | 1 | 0
Not completed — Failed to return | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Population (SAP) comprised all participants who received at least one dose of study medication. The SAP was used for all efficacy and safety analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.8 (0.45) | 4.0 (1.08) | 3.1 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Plasma Trough Concentrations (Ctrough) for Saquinavir
Description: Plasma trough concentration is the average steady state concentration prior to morning and evening dose. Ctrough of Saquinavir was normalized to a dose of 50 mg/kg.
Time Frame: Pre-dose at Weeks 8, 12, 24.
Population: The pharmacokinetics Analysis Population (PKP) comprised all the participants from whom blood samples for pharmacokinetic analysis were collected. Participants could be excluded from the PKP if no reliable PK parameters could be determined or if justified by circumstances (e.g. vomiting after drug administration) and in agreement with the sponsor.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 5 | 13
ng/mL | 645 (536) | 1860 (1060)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to Twelve Hours (AUC0-12h) for Saquinavir
Description: The area under the plasma concentration-time curve from time zero to twelve hours (AUC0-12h) is area under the plasma concentration-time curve from time zero through actual tlast. The area under the plasma concentration-time curve from time zero to twelve hours of saquinavir was normalized to a dose of 50 mg/kg.
Time Frame: Pre-dose and 3, 4, 8, 12 hours (post-dose) on Day 14 (± 2 days), or Day 28(+ 2 days) for patients switching from an Non-nucleoside reverse transcriptase inhibitor [NNRTI] containing regimen).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 5 | 13
h*ug/mL | 18.7 (20.0) | 38 (18.1)

3. Primary Outcome: Incidence of Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes
Time Frame: From Baseline (Day 1) till Week 48 and Follow-up (Week 52)
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Total: Participants received saquinavir at a dose of 50 mg/Kg BID and ritonavir at a dose of 3 mg/kg BID for body weight from 5 to < 15 kg, 2.5 mg/kg BID for body weight from 15 to 40 kg and 100 mg BID for body weight > 40 kg plus >= 2 background ARVs. After 14 days of treatment (or Day 28 for participants switching from an NNRTI containing regimen), saquinavir and ritonavir dose adjustments were made within the age group or for individual participants as deemed appropriate. The highest dose for saquinavir/ritonavir that was to be administered was not to exceed 1000 mg/100 mg BID. Participants received treatment for 48 weeks.
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
participants
  Any serious adverse events | 1 | 2 | 3
  Any non-serious adverse events | 5 | 9 | 14

4. Primary Outcome: Change In Hematocrit From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: The Safety Analysis Population comprised all patients who received at least one dose of study medication. The SAP was used for all efficacy and safety analyses.
Measure: Mean (Standard Deviation); unit: fraction
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
fraction
  Change from Baseline at Week 24 (n= 4, 13, 17) | 0.01 (0.011) | -0 (0.03) | -0 (0.027)
  Change from Baseline at Week 48 (n= 4, 13, 17) | 0.03 (0.037) | -0.01 (0.044) | 0 (0.044)

5. Secondary Outcome: Plasma Trough Concentrations (Ctrough) for Ritonavir
Description: Plasma trough concentration is the average steady state concentration prior to morning and evening dose. Ctrough of Ritonavir was normalized to a dose of 100 mg/kg.
Time Frame: Pre-dose at Weeks 8, 12, 24
Population: The PKP population comprised all the participants from whom blood samples for pharmacokinetic analysis were collected. Participants could be excluded from the PKP if no reliable PK parameters could be determined or if justified by circumstances (e.g. vomiting after drug administration) and in agreement with the sponsor.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 5 | 13
ng/mL | 577 (366) | 995 (548)

6. Secondary Outcome: Maximum Observed Concentration (Cmax) for Saquinavir and Ritonavir
Description: The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration. Cmax was normalized to a dose of 50 mg/kg for Saquinavir and100 mg/kg for Ritonavir.
Time Frame: Pre-dose and 3, 4, 8, 12 hours (post-dose) on Day 14 (± 2 days), or Day 28(+ 2 days) for patients switching from an NNRTI containing regimen and at Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 5 | 13
ng/mL
  Saquinavir | 2910 (3110) | 5570 (2780)
  Ritonavir | 2050 (1270) | 3370 (2020)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to Twelve Hours (AUC0-12h) for Ritonavir
Description: The area under the plasma concentration-time curve from time zero to twelve hours (AUC0-12h) is area under the plasma concentration-time curve from time zero through actual tlast. The area under the plasma concentration-time curve from time zero to twelve hours of ritonasvir was normalized to a dose of 100 mg/kg.
Time Frame: Pre-dose and 3, 4, 8, 12 hours (post-dose) on Day 14 (± 2 days), or Day 28(+ 2 days) for patients switching from an NNRTI containing regimen).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 5 | 13
h*ug/mL | 13.6 (8.18) | 21.8 (11.6)

8. Secondary Outcome: Change From Baseline in Mean Human Immunodeficiency Virus Viral Load
Description: Change from baseline in plasma HIV-1 RNA was derived as Change from baseline = Log10 (HIV-1 RNA at week x) - Log10 (HIV-1 RNA at baseline)
Time Frame: Baseline (Day 1), Weeks 8, 12, 24, 36, and 48 (or upon premature discontinuation); a baseline collection was made if there was not already a value available taken within the previous 4 weeks.
Population: The Safety Analysis Population (SAP) comprised all patients who received at least one dose of study medication. The SAP was used for all efficacy and safety analyses.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
log10 copies/mL
  Change from Baseline at Week 24 (n= 3, 13, 16) | -0.75 (1.48) | -1.81 (1.57) | -1.61 (1.57)
  Change from Baseline at Week 48 (n= 3, 13, 16) | -1.27 (1.01) | -1.39 (1.53) | -1.36 (1.42)

9. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV) -Ribonucleic Acid (RNA) <400 Copies/mL
Description: The number of participants with HIV-1 RNA results <400 copies/mL were reported
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
participants
  Baseline (n= 5, 13, 18) | 1 | 5 | 6
  Week 24 (n= 3, 13, 16) | 2 | 13 | 15
  Week 48 (n= 3, 13, 16) | 2 | 11 | 13

10. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV) -Ribonucleic Acid (RNA) <50 Copies/mL
Description: The number of participants with HIV-1 RNA results <50 copies/mL were reported.
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
participants
  Baseline (n= 5, 13, 18) | 0 | 4 | 4
  Week 24 (n= 3, 13, 16) | 2 | 11 | 13
  Week 48 (n= 3, 13, 16) | 2 | 9 | 11

11. Secondary Outcome: Number of Participants With >1 Log Decrease From Baseline in Human Immunodeficiency Virus (HIV) -Ribonucleic Acid (RNA )
Description: The number of participants experiencing a greater than 1 log drop from baseline (day 1) (log 10 transformed) were reported
Time Frame: From Week 8 till Week 48
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
participants
  Week 8 (n= 4, 12, 16) | 1 | 7 | 8
  Week 24 (n= 3, 13, 16) | 1 | 8 | 9
  Week 48 (n= 3, 13, 16) | 1 | 7 | 8

12. Secondary Outcome: Number of Participants With Virological Failure
Description: Virological failure was defined as: viral load >= 400 copies/mL on two consecutive occasions (missing visits was assumed to be above 400 copies/mL). The number of participants classified as virological failure by Age Group and viral load (≤ 10,000 copies, >10,000 copies) were presented.
Time Frame: From Week 12 till Week 48
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
participants
  VF at Week 12 (n= 5, 13, 18) | 2 | 1 | 3
  VF at Week 24 (n= 5, 13, 18) | 2 | 0 | 2
  VF at Week 48 (n= 5, 13, 18) | 3 | 1 | 4
  HIV-RNA <= 10,000 copies/mL at Wk 12 (n= 3, 6, 9) | 1 | 0 | 1
  HIV-RNA <= 10,000 copies/mL at Wk 24 (n= 3, 6, 9) | 1 | 0 | 1
  HIV-RNA <= 10,000 copies/mL at Wk 48 (n= 3, 6, 9) | 2 | 0 | 2
  HIV-RNA >10,000 copies/mL at Week 12 (n= 2, 7, 9) | 1 | 1 | 2
  HIV-RNA >10,000 copies/mL at Week 24 (n= 2, 7, 9) | 1 | 0 | 1
  HIV-RNA >10,000 copies/mL at Week 48 (n= 2, 7, 9) | 1 | 1 | 2

13. Secondary Outcome: Change From Baseline in Cluster Differentiation Antigen 4 (CD4) Lymphocyte Count
Description: Change from Baseline in CD4+ lymphocyte count at 24 weeks and 48 weeks were presented by age group. Change from baseline in CD4+ lymphocyte count was derived as follows: Change from baseline = (CD4+ count at week 24/48) - (CD4+ count at baseline). A baseline collection was made if there was not already a value available taken within the previous 4 weeks. Baseline was on Day 1.
Time Frame: Baseline (Day 1), Weeks 8, 12, 24, 36, and 48 or upon premature discontinuation
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: count/uL
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
count/uL
  Change from Baseline at Week 24 (n= 3, 12, 15) | 94.90 (643.28) | -34.53 (821.31) | -8.65 (769.41)
  Change from Baseline at Week 48 (n= 3, 12, 15) | -50.07 (1013.23) | 126.11 (528.49) | 90.87 (609.46)

14. Secondary Outcome: Change From Baseline in Cluster Differentiation Antigen 8 (CD8) Lymphocyte Count
Description: Change from baseline in CD8+ lymphocyte count at 24 weeks and 48 weeks were presented by age group. Change from baseline in CD8+ lymphocyte count was derived as follows: Change from baseline = (CD8+ count at week 24/48) - (CD8+ count at baseline). A baseline collection was made if there was not already a value available taken within the previous 4 weeks. Baseline was on Day 1.
Time Frame: Baseline (Day 1), Weeks 8, 12, 24, 36, and 48 or upon premature discontinuation
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: count/uL
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
count/uL
  Change from Baseline at Week 24 (n= 3, 12, 15) | -200.49 (161.05) | -3.50 (790.86) | -42.90 (708.37)
  Change from Baseline at Week 48 (n= 3, 12, 15) | -92.07 (455.23) | 40.52 (641.27) | 14.00 (596.43)

15. Primary Outcome: Change In Hemoglobin, Total Protein And Total Albumin From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
g/L
  Hemoglobin, Change from BL at Wk 24 (n= 4, 13, 17) | -0 (3.3) | 1 (12.1) | 1 (10.6)
  Hemoglobin, Change from BL at Wk 48 (n= 4, 13, 17) | 6 (11.8) | 0 (14.4) | 2 (13.7)
  Total Protein, Change from BL at Wk 24 (n=4,13,17) | -4 (6.0) | 2 (12.6) | 0 (11.5)
  Total Protein, Change from BL at Wk 48 (n=4,13,17) | -5 (5.7) | -0 (14.3) | -1 (12.8)
  Total Albumin, Change from BL at Wk 24 (n=4,13,17) | 0.5 (5.41) | 5 (7.68) | 4 (7.32)
  Total Albumin, Change from BL at Wk 48 (n=4,13,17) | 1.3 (2.29) | 4 (8.7) | 3.4 (7.7)

16. Primary Outcome: Change In White Blood Cell (WBC), Platelet, Basophil, Lymphocyte, Monocyte, Neutrophil And Eosinophil Cell Counts From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10*9/L
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
10*9/L
  WBC, Change from BL at Wk 24 (n= 4,13,17) | -3 (2.31) | -1 (4.35) | -1.5 (4.0)
  WBC, Change from BL at Wk 48 (n= 4,13,17) | -2.1 (1.72) | -0.9 (4.38) | -1.2 (3.9)
  Platelet, Change from BL at Wk 24 (n= 4,13,17) | -119 (93.4) | 24 (148.9) | -9 (148.9)
  Platelet, Change from BL at Wk 48 (n= 4,13,17) | -50 (130.4) | -2 (118.9) | -13 (119.3)
  Basophil, Change from BL at Wk 24 (n=4 ,13,17) | -0.02 (0.028) | 0 (0.031) | -0.01 (0.031)
  Basophil, Change from BL at Wk 48 (n=4 ,13,17) | -0 (0.03) | -0.01 (0.029) | -0.01 (0.028)
  Lymphocyte, Change from BL at Wk 24 (n=2, 2, 4) | -0.9 (0.3) | -1.1 (1.20) | -1 (0.72)
  Lymphocyte, Change from BL at Wk 48 (n= 2, 2, 4) | -1.5 (0.29) | -0.7 (1.05) | -1.1 (0.76)
  Monocyte, Change from BL at Wk 24 (n= ,13,17) | -0.41 (0.295) | -0.01 (0.361) | -0.11 (0.379)
  Monocyte, Change from BL at Wk 48 (n= ,13,17) | -0.21 (0.179) | -0.05 (0.384) | -0.09 (0.348)
  Neutrophil, Change from BL at Wk 24 (n=2, 2, 4) | -1.4 (0.33) | -2.8 (1.87) | -2.1 (1.36)
  Neutrophil, Change from BL at Wk 48 (n= 2, 2, 4) | -1.7 (1.15) | -1.6 (2.55) | -1.6 (1.62)
  Eosinophil, Change from BL at Wk 24 (n=2, 2, 4) | -0 (0.2) | -0 (0.1) | -0 (0.1)
  Eosinophil, Change from BL at Wk 48 (n= 2, 2, 4) | -0 (0.2) | 0 (1.1) | 0 (0.7)

17. Primary Outcome: Change In Red Blood Cell (RBC) Counts From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10*12/L
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
10*12/L
  RBC,Change from Baseline at Week 24 (n= 4, 13, 17) | -0.18 (0.227) | -0.07 (0.673) | -0.1 (0.593)
  RBC,Change from Baseline at Week 48 (n= 4, 13, 17) | 0.02 (0.125) | -0.16 (0.74) | -0.12 (0.648)

18. Primary Outcome: Change In Creatine Kinase (CK), Serum Glutamic Oxaloacetic Transaminase (SGOT), Alkaline Phosphatase (ALP), Serum Glutamic-Pyruvic Transaminase (SGPT), Gamma-Glutamyl Transferase (GGT) Counts From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
U/L
  CK, Change from Baseline at Week 24 (n= 3, 3, 16) | 112 (112.0) | -12 (115.9) | 11 (122.2)
  CK, Change from Baseline at Week 48 (n= 3, 3, 16) | 257 (244.8) | -7 (84) | 43 (158)
  SGOT, Change from Baseline at Week 24 (n= 4,13,17) | -0 (1.5) | -0 (8.2) | -0 (7.1)
  SGOT, Change from Baseline at Week 48 (n= 4,13,17) | -1 (7.8) | -0 (6.9) | -0 (6.8)
  ALP, Change from Baseline at Week 24 (n=4, 12, 16) | 10 (29.8) | 26 (23.2) | 22 (24.9)
  ALP, Change from Baseline at Week 48 (n=4, 12, 16) | 47 (87.6) | 36 (26.5) | 39 (45.6)
  SGPT, Change from Baseline at Week 24 (n=4,13,17) | -9 (15.3) | -2 (13.6) | -4 (13.8)
  SGPT, Change from Baseline at Week 48 (n=4,13,17) | -2 (13.4) | -3 (12.1) | -3 (12)
  GGT, Change from Baseline at Week 24 (n=4, 13, 17) | 5 (4.7) | -7 (18.7) | -4 (17.1)
  GGT, Change from Baseline at Week 48 (n=4, 13, 17) | 5 (2.1) | -5 (18.5) | -2 (16.7)

19. Primary Outcome: Change In Total Bilirubin, Creatinine, Uric Acid From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
umol/L
  Total Bilirubin-Change from BL at Wk 24(n=4,12,16) | 2 (2.8) | 2 (5.5) | 2 (4.9)
  Total Bilirubin-Change from BL at Wk 48(n=4,12,16) | 1 (1.1) | 2 (6.9) | 1 (5.9)
  Cretainine- Change from BL at Wk 24 (n=4, 13,17) | -2 (6.7) | 3 (10) | 2 (9.5)
  Cretainine- Change from BL at Wk 48 (n=4, 13,17) | 3 (10.7) | 5 (9.2) | 5 (9.3)
  Uric acid- Change from BL at Wk 24 (n=4, 13,17) | -27 (54.3) | 68 (55.1) | 46 (67.6)
  Uric acid- Change from BL at Wk 48 (n=3,13,16) | -42 (108.4) | 61 (63.5) | 41 (80.6)

20. Primary Outcome: Change In Blood Urea Nitrogen (BUN), Low Density Lipoprotein (LDL) Cholesterol, High Density Lipoprotein (HDL Cholesterol), Triglycerides, Calcium, Potassium, Sodium, Chloride, Phosphate, Fasting Glucose From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
mmol/L
  BUN,Change from Baseline at Week 24 (n= 3, 13, 16) | -1.5 (2.78) | 1 (2.2) | 0.5 (2.43)
  BUN,Change from Baseline at Week 48 (n= 3, 13, 16) | 0.4 (0.66) | 1.1 (2.0) | 0.9 (1.82)
  LDL,Change from Baseline at Week 24 (n= 3, 13, 16) | 0.21 (0.237) | 0.21 (1.389) | 0.21 (1.245)
  LDL,Change from Baseline at Week 48 (n= 3, 13, 16) | 0.23 (0.596) | -0.11 (1.038) | -0.04 (0.963)
  HDL,Change from Baseline at Week 24 (n= 3, 13, 16) | 0.21 (0.202) | 0.13 (0.369) | 0.15 (0.34)
  HDL,Change from Baseline at Week 48 (n= 3, 13, 16) | 0.41 (0.233) | 0.17 (0.387) | 0.21 (0.37)
  Triglyceride,Change from BL at Wk 24 (n=4,13, 17) | -0.28 (0.597) | -0.19 (1.376) | -0.21 (1.22)
  Triglyceride,Change from BL at Wk 48 (n=4,13, 17) | -0.19 (0.496) | -0.15 (1.558) | -0.16 (1.366)
  Calcium,Change from BL at Wk 24 (n=2, 12, 14) | -0.15 (0.04) | 0.15 (0.17) | 0.11 (0.19)
  Calcium,Change from BL at Wk 48 (n=2, 12, 14) | -0.16 (0.09) | 0.09 (0.17) | 0.06 (0.18)
  Potassium,Change from BL at Wk 24 (n=4,13, 17) | -0.1 (0.16) | -0.3 (0.63) | -0.2 (0.56)
  Potassium,Change from BL at Wk 48 (n=4,13, 17) | 0.2 (0.59) | -0.2 (0.54) | -0.1 (0.57)
  Sodium,Change from BL at Wk 24 (n=4,13, 17) | 2 (1.3) | -1 (2.3) | -0 (2.3)
  Sodium,Change from BL at Wk 48 (n=4,13, 17) | 1 (2.2) | -1 (3.8) | -0 (3.5)
  Chloride,Change from BL at Wk 24 (n=4,13, 17) | -1 (2.8) | -2 (4.2) | -2 (3.9)
  Chloride,Change from BL at Wk 48 (n=4,13, 17) | 1 (1.3) | -2 (3.6) | -1 (3.3)
  Phosphate,Change from BL at Wk 24 (n=2, 12, 14) | -0.02 (0.114) | 0.17 (0.188) | 0.14 (0.188)
  Phosphate,Change from BL at Wk 48 (n=2, 13, 15) | -0.26 (0.0) | 0.12 (0.212) | 0.07 (0.237)
  Fasting Glucose,Change from BL at Wk 24(n=4,13,17) | -0.26 (0.963) | 0.02 (1.253) | -0.05 (1.169)
  Fasting Glucose,Change from BL at Wk 48(n=4,13,17) | -0.07 (0.857) | 0.14 (1.537) | 0.09 (1.385)

21. Primary Outcome: Change In Hematuria, Glycosuria And Proteinuria From Baseline
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: [0 to 4+]
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 13 | 18
[0 to 4+]
  Hematuria-Change from BL at Wk 24 (n= 1, 2, 3) | 0 (0) | 0 (0) | 0 (0)
  Hematuria-Change from BL at Wk 48 (n= 1, 2, 3) | 0 (0) | 0 (0) | 0 (0)
  Glycosuria-Change from BL at Wk 24 (n= 1, 2, 3) | 0 (0) | 0 (0) | 0 (0)
  Glycosuria-Change from BL at Wk 48 (n= 1, 2, 3) | 0 (0) | 0 (0) | 0 (0)
  Proteinuria-Change from BL at Wk 24 (n= 1, 2, 3) | 0 (0) | 0 (0) | 0 (0)
  Proteinuria-Change from BL at Wk 48 (n= 1, 2, 3) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Up to 56 weeks
Description: Serious adverse events and non-serious adverse events are reported in Safety Population Set.
Arm/Group | Group A | Group B | Total
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/13 | 3/18
Other Adverse Events (participants affected / at risk) | 5/5 | 9/13 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=5) | Group B (N=13) | Total (N=18)
Pneumonia (Infections and infestations) | 1 | 1 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=5) | Group B (N=13) | Total (N=18)
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 2 | 2
Impetigo (Infections and infestations) | 0 | 1 | 1
Otitis Media (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Giardiasis (Infections and infestations) | 1 | 0 | 1
Herpangina (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Otitis Media Acute (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pyoderma (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Toxocariasis (Infections and infestations) | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3
Dental Caries (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Gait Disturbance (General disorders) | 1 | 0 | 1
Weight Decreased (Investigations) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Enuresis (Renal and urinary disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.